CLINICAL TRIAL: NCT06853158
Title: MULTIsite Feasibility of MUSIc Therapy to Address Quality Of Life in Sickle Cell Disease (MULTI-MUSIQOLS)
Brief Title: MULTIsite Feasibility of MUSIc Therapy to Address Quality Of Life in Sickle Cell Disease
Acronym: MULTI-MUSIQOLS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of California, San Francisco (Other); Case Western Reserve University (Other); Prisma Health-Upstate (Other); University of Massachusetts Chan Medical School, Worcester (Unknown)
Responsible Party: Principal Investigator, Jeffrey Dusek, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 5448; 7R01AT012508-02 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: feasibility, music therapy, QoL, Sickle cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Type/design of trial This is a multi-site, multi-visit feasibility RCT of three wellbeing interventions among patients aged 14 and older with SCD.
  Specific unit(s) of assignment and unit(s) of observation
  The unit of assignment is at the patient level. Specifically, patients with SCD enrolled from SCD centers will be randomly assigned to either InMT, HybMT or HybHE. The unit of observation is the patient.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Multiple Principal Investigators (Drs. Dusek and Jenerette) will be unaware of treatment assignment as will the site PIs. The statisticians who will be assessing feasibility will also be unaware of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- InMT (Experimental): Participants in the InMT will receive 6 in-person MT sessions at the SCD center main campus, satellite campus, or another location preferred by the participant (e.g., community center).
  Interventions: Behavioral: Music therapy
- HybMT (Experimental): Individuals randomized to Hybrid MT will receive 1 in-person MT session at the SCD center main campus, satellite campus, or another location preferred by the participant (e.g., community center) and 5 virtual MT sessions over secure telehealth platform (e.g. Zoom Health Professional).
  Interventions: Behavioral: Music therapy
- HybHE (Active Comparator): Participants in the HybHE condition will receive 1 in-person health education session at the SCD center main campus, satellite campus, or another location preferred by the participant (e.g., community center) and 5 virtual sessions over secure telehealth platform (e.g. Zoom Health Professional).
  Interventions: Other: Health education

INTERVENTIONS:
Behavioral: Music therapy — Participants in the 2 experimental MT conditions (In person MT (InMT) or hybrid (inperson.virtual (HybMT) will receive 6 MT sessions over 6 weeks. Each MT session will last no longer than one hour. This 6-week treatment period may be extended to up to 8 weeks if a scheduling conflict prevents a participant from receiving the 6 MT sessions over 6 consecutive weeks.
  Arms: HybMT; InMT
Other: Health education — The content for the HybHE control was adapted from Project PEEP: Patients Empowered and Educated Providers. The Sickle Cell Community Consortium developed Project PEEP with a grant from Global Blood Therapeutics. Project PEEP addresses unmet needs directly identified and prioritized by a collective of patients with SCD, caregivers, and community-based organizations. The objective is to provide the tools and resources to improve communication and increase positive patient-provider interactions to receive quality, timely care. For the proposed study, we will use modules from the curriculum developed for patients living with SCD.
  Arms: HybHE

SUMMARY:
This is a multi-site, multi-visit feasibility RCT of music therapy (MT) among adolescent and adult patients (aged 14 and older) with sickle cell disease (SCD).

Subjects will be randomized into one of three groups, either (1) 6 visits of in- person MT (InMT:); (2) 1 visit of in-person MT and 5 visits of virtual MT (HybMT); or (3) 1 visit of in-person health education and 5 visits of virtual health education (HybHE).

Cohorts of 15 participants (10 at site 1 and 5 site 2) will be recruited each quarter for 6 quarters to reach 90 participants. Cohorts will maintain a semi-structured recruitment, consenting, assessment, and intervention schedule.

The primary objective of the study is to examine the feasibility of study. This is defined by 6 metrics: (1) completeness of data collection, (2) participant screening, (3) participant recruitment, (4) participant retention, (5) Individual attendance and (6) Home practice. A final determination of "feasibility" for the study will be met if any 4 of the 6 metrics described above are met.

This study will also include a secondary objective of conducting qualitative interviews to assess feasibility of implementation.

DETAILED DESCRIPTION:
The objectives of this study are to (1) conduct a feasibility randomized control trial (RCT), to examine the data collection processes, and intervention (in-person music therapy [InMT], hybrid MT [HybMT], and hybrid health education [HybHE]) implementation overall and across 2 sites (University Hospitals/Case Western Reserve University [site 1] and Prisma Health/University of South Carolina [site 2]); and (2) evaluate the implementation of the InMT, HybMT, and HybHE interventions using both quantitative data (study records, stakeholder surveys) and qualitative data (interviews).

Three wellbeing programs for individuals with SCD will be compared: (1) InMT, (2) HybMT, and (3) HybHE. Each intervention includes 6 sessions. The treatment period for each group will be 6 to 8 weeks. Each weekly session will last up to one hour in all arms of the study. MT sessions in the InMT and HybMT arms will include the topics of SCD education and MT rationale, breathing exercises, relaxation, imagery, music making, and review and creation of a coping plan for future challenges. The HybHE group will use an adapted version of Project Patients Empowered and Educated Providers (PEEP). Covered topics include: science of SCD, identifying barriers in the Emergency Department, tools for navigating the healthcare system, healthcare based communication, and review and planning for future challenges.

Semi-structured qualitative interview topics will focus on participants' perceptions of the interventions, perceived benefits and burdens of the interventions, and other barriers and facilitators to in-person and hybrid delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged >=14 years old
2. Have a diagnosis of SCD present in their electronic health record (EHR);
3. Meet Analgesic, Anesthetic, and Addiction Clinical Trial Translations Innovations Opportunities and Networks-American Pain Society Pain Taxonomy (AAPT) criteria for chronic SCD pain which includes:

3a. A diagnosis of SCD confirmed by laboratory testing (present in EHR per eligibility criteria 2)

3b. Reports of ongoing pain present on most days over the past 6 months either in a single location or in multiple locations (to be obtained at screening)

3c. Displaying at least one of the following signs on clinical exam (to be obtained from providers' clinical notes in the EHR

* Palpation of the region of reported pain elicits focal pain or tenderness;
* Movement of the region of reported pain elicits focal pain;
* Decreased range of motion or weakness in the region of reported pain;
* Evidence of skin ulcer in the region of reported pain;
* Evidence of hepatobiliary or splenic imaging abnormalities (e.g., splenic infarct, chronic pancreatitis) consistent with the region of reported pain; or
* Evidence of imaging abnormalities consistent with bone infarction or avascular necrosis in the region of reported;

  3d. There is no other diagnosis that better explains the signs and symptoms (to be obtained from providers following referral and pre-screening)

  4. Be able to speak and understand English;

  5. Have an email address and access to mobile device with a functioning data plan

  6. Reporting that pain interfered with daily activities at least 1-2 days in the past week.

Exclusion Criteria:

1. Have a significant visual, hearing, or cognitive impairment
2. Have previously participated in the MUSIQOLS single-site pilot study at University Hospitals in 2018
3. Are currently engaging in mind-body therapies under the supervision of a healthcare professional specifically for pain management
4. Have a planned major medical event in the next 14 weeks such as (but not limited to) childbirth, orthopedic surgery, gene therapy, or stem cell transplant (These criteria do not include blood transfusions, exchange transfusions, or other pharmacologic pain treatment).

Qualitative interviews will be conducted with ~24 participants who received the interventions (with equal numbers across the InMT, HybMT and HybHE groups). Participants will be purposively sampled to include equal distribution across sites in proportion to recruitment.

Stakeholder surveys and qualitative interviews will be conducted among ~20 relevant staff stakeholders (~10 per site), including healthcare providers & staff, music therapists and HybHE interventionists.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Multi Musiqols Overall Feasibility (achieving 4/6 of the secondary outcomes). | through study completion, an average of 1 year
  There are 6 feasibility metrics: (1) Data quality (90%), (2) Screening rate (35%), (3) Recruitment rate (90%), (4) Retention rate (70%), (5) Individual attendance (70%) and (6) Home practice (70%). A final determination of "feasibility" for the study will be met if any 4 of the 6 metrics are met.

SECONDARY OUTCOMES:
Data quality and completeness (90% goal) | through study completion, an average of 1 year
  This variable is described as being the number of data elements that are correctly completed in the Multi Musiqols REDCap project. The feasibility goal is 90%
Successful Screening Rate of Enrolled Individuals (35% goal) | At enrollment
  The screening rate as those who were enrolled (i.e., provide written informed consent) divided by those approached for the study who met eligibility criteria. The feasibility goal is 35%.
Successful Recruitment of Participants into the Study (90% goal) | At Enrollment
  This translates into randomizing 90% participants who provided written informed consent
Successful Retention of Participants (70% goal) | through study completion, an average of 1 year
  This metric is defined as the number of participants retained until the final survey time point (6-week follow-up) divided by the number of randomized participants.
Successful Individual Attendance of Study Sessions (70% goal) | through study completion, an average of 1 year
  We will consider individual attendance to be acceptable if a given participant attends 4 of 6 sessions in 8 weeks. These 4 sessions must include the first session and any 3 out of the 4 sessions between sessions 2-5. Individual session attendance will be deemed complete if the participant attends 2/3 of the session including (1) the introduction (discussing experience with the MT or HybHE exercise over previous week, providing education on rationale for intervention); (2) setting of the agenda; and (3) the main intervention (e.g., co-creating the music for the intervention, customizing the place and imagery to participants' preferences, experiencing and recording the intervention).
Successful Individual Home Practice (70%) | At 6 week follow-up
  If a given participant practices intervention exercises at least once per week, this will be coded as engaging in the minimum dose of home practice.

OTHER OUTCOMES:
Participant Satisfaction Question 1 | At 6 week follow-up
  Enrolled participants will be asked "How satisfied are you with how your pain was managed during your participation in the study" on the 5-point Likert scale (1-strongly dissatisfied-5-very satisfied). Qu 1 will be asked at treatment completion and at 6-week follow up.
Participant Satisfaction Question 2 | At 6 week follow-up
  Enrolled participants will be asked ""Overall how satisfied are you with your treatment during your study participation?" on the same 5-point Likert Scale. Qu 2 will be asked at treatment completion and at 6-week follow up.
Provider Satisfaction Question 1 | through study completion, an average of 1 year
  Providers will be asked: "To what degree do you view the InMT, HybMT or HybHE intervention as useful or suitable for this population?" (1- very inappropriate-5-very appropriate).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery A Dusek, PhD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - UH Seidman Cancer Center Adult SCD Clinic or UH Rainbow Babies and Children's Hospital Sickle Cell Anemia Center, Cleveland, Ohio
  - Prisma Health Lifespan Comprehensive SCD Program, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT06853158/Prot_SAP_001.pdf